CLINICAL TRIAL: NCT01049581
Title: Effects of Pediatric Aquatic Therapy in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 981947B
Record Dates: First submitted 2010-01-04; First posted 2010-01-14 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Spastic Cerebral Palsy
Keywords: Gross motor function performance; pediatric aquatic therapy; spastic cerebral palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Aquatic Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pediatric aquatic therapy (Experimental): The children of the PAT group participated in a 1 hour/time, twice-per-week, 12-week, PAT program in addition to conventional rehabilitation programs
  Interventions: Procedure: aquatic therapy
- conventional therapy (No Intervention): The children included in the control group continued with their original rehabilitation programs

INTERVENTIONS:
Procedure: aquatic therapy — two hours per week, one hour per time, total 12 weeks
  Other Names: physical therapy
  Arms: pediatric aquatic therapy

SUMMARY:
Aquatic intervention had been applied in children with neuromotor impairment for years, yet there has been little progress toward objective identifications of therapy goals, interventions, and outcomes. Thus, we attempt to design aquatic intervention activity for children with cerebral palsy to evaluate the effect of hydrotherapy.

Purpose:

To evaluate the effects of pediatric aquatic therapy on motor performance, daily activity and social participation in children with spastic cerebral palsy.

Method:

The study enrolled 27 children with spastic cerebral palsy aged from 4 to 12 years old.These children were dived into two groups: traditional rehabilitation therapy (control group), and hospital based pediatric aquatic therapy program. We evaluate the motor performance, daily activity and social participation before and after the intervention and compared the difference in improvement between groups. The measurements include modified Ashworth score, Gross Motor Function Measure (GMFM -66), Vineland Adaptive Behavior Scale (VABS) , and Cerebral Palsy Quality of Life Questionnaire for Children (CPQOL).

Expect effect:

We suppose pediatric aquatic therapy in spastic cerebral palsy children could improve motor function and daily activity.Children could improve self-esteem and we hypothesize this could improve social participation.

DETAILED DESCRIPTION:
* We conducted a well-designed study to investigate the effectiveness of PAT on motor function, activities of daily living (ADL),and health related quality of life(HRQOL) perspectives for children with CP.
* A convenience sample of 27 children was recruited for the study from the outpatient clinics of the Department of Physical Medicine and Rehabilitation of two tertiary hospitals: Chang Gung Memorial Hospital and Taipei Veterans General Hospital.
* The study was designed as a single blinded, prospective, case control study.
* The pediatric aquatic therapy group got more improvementon motor performance measured by GMFM-66.

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed as cerebral palsy, spastic type
2. Gross Motor Functional Classification (GMFCS) level II-IV
3. Age: 4-12 y/o
4. Informed consent by parents
5. Modified Ashworth score 2 or3
6. If participant history of epilepsy ,well controlled by medication

Exclusion Criteria:

1. History of psychiatric diseases
2. Poor controlled epilepsy
3. Received botox injection or surgery in recent three months
4. Children diagnosed as attention deficit hyperactivity disorder(ADHD) or autism
5. Severe mental retardation
6. Active infection (Body temperature > 100°F)
7. Communication problems
8. Bowel incontinence
9. Bladder incontinence
10. Severe cardiovascular disease
11. Infectious skin conditions and open wound
12. Nasogastric tubes or gastrostomy tubes
13. Colostomy ,urostomy or ileostomy bags
14. Acute orthopedic injury with pain and instability
15. Diabetes
16. Chlorine sensitivity
17. Latex allergies
18. Tracheostomy

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ChiaLing Chen, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A convenience sample of 27 children was recruited for the study from the outpatient clinics of the Department of Physical Medicine and Rehabilitation of two tertiary hospitals: Chang Gung Memorial Hospital and Taipei Veterans General Hospital.
Pre-assignment Details: Exclusion * Children receiving botulinum toxin injection or surgery within 3 months * psychiatric diseases or communication disorders * poorly controlled epilepsy, * skin problems such as open wound
Groups:
- Pediatric Aquatic Therapy Group: *Children diagnosed with cerebral palsy, spastic type,*4 to 12 years of age,*Goss Motor Functional Classification System (GMFCS) level I-IV,participate the pediatric aquatic therapy according to preference
- Conventional Therapy Group: *Children diagnosed with cerebral palsy, spastic type,*4 to 12 years of age,*Goss Motor Functional Classification System (GMFCS) level I-IV,participate the conventional therapy according to preference
Period: Overall Study
Arm/Group | Pediatric Aquatic Therapy Group | Conventional Therapy Group
Started | 13 | 14
Completed | 11 | 13
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pediatric Aquatic Therapy Group: The participants were classified into two groups the pediatric aquatic therapy group according the their preference. The children of the PAT group participated in a 1 hour/time, twice-per-week, 12-week, PAT program in addition to conventional rehabilitation programs.
- Conventional Therapy Group: The participants were classified into the control (conventional therapy) group according to preference. The children included in the control group continued with their original rehabilitation programs.
- Total: Total of all reporting groups
Arm/Group | Pediatric Aquatic Therapy Group | Conventional Therapy Group | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 14 | 27
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7 (3) | 6 (2.5) | 7 (0.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  Taiwan | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Unit on Gross Motor Function Measure Scale (GMFM)
Description: The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy. The scoring key is meant to be a general guideline. However, most of the items have specific descriptors for each score. It is imperative that the guidelines contained in the manual be used for scoring each item. The score ranges from 0 to 100 and the higher represent the better gross motor function in children with cerebral palsy
Time Frame: 3 months
Population: complete the study and examination
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pediatric Aquatic Therapy: 13 children diagnosed as spastic cerebral palsy participate to pediatric aquatic therapy according preference and finally 11 children complete the study
- Conventional Therapy: Initially 14 children diagnosed as spastic cerebral palsy participate conventional therapy according to preference and 13 children complete the study
Arm/Group | Pediatric Aquatic Therapy | Conventional Therapy
Number analyzed (Participants) | 11 | 13
units on a scale | 5.12 (4.5) | 2.00 (2.7)
Statistical Analysis 1: Comparison: Pediatric Aquatic Therapy vs Conventional Therapy; null hypothesis : there is no difference in gross motor performance in pediatric aquatic therapy group and conventional therapy group; Test type: Non-Inferiority or Equivalence — ANCOVA was used and the result reveled (F1, 17 = 7.565, η2= 0.308, p = 0.007); p = 0.007, ANCOVA

2. Secondary Outcome: Daily Living Subscale of Vineland Adaptive Behavior Scale
Description: Vineland Adaptive Behavior scale was developed by Sara et al at 1984 and was used to measure adaptive and maladaptive behavior in children age form 3-12 years-old. The daily living subscale range from 0 to 198 and the higher the score represent the better captive behavior.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pediatric Aquatic Therapy: 13 children diagnosed as spastic type cerebral palsy participate pediatric auqatic therapy and 11 children finish the study,each of them fulfill the the questionnaire before and after the intervention
- Conventional Therapy: 14 children diagnosed as spastic type cerebral palsy participate conventional therapy and 13 children finish the study,each of them fulfill the the questionnaire before and after the intervention
Arm/Group | Pediatric Aquatic Therapy | Conventional Therapy
Number analyzed (Participants) | 11 | 13
units on a scale | 81.8 (48.9) | 92.1 (38.5)
Statistical Analysis 1: Comparison: Pediatric Aquatic Therapy; We hypothesize that Children with CP receiving PAT would have better outcomes in motor function and translate to ADL; Test type: Non-Inferiority or Equivalence — ANCOVA : p value 0.393; p = 0.393, ANCOVA — Effect Size η2 0.023; F1,17= 0.380; Mean Difference (Net) = 1.762

3. Secondary Outcome: Subscale on Cerebral Palsy Quality of Life Questionnaire for Children
Description: This questionnaire was developed for Children and was a condition-specific quality of life (QOL) questionnaire for children with cerebral palsy aged 4 to 12 years. It contains social , functioning, participation , emotional ,access, pain and disability, and family health components. Participation is the main component in this study. This sub score ranges from 0 to 81 , higher scores represent better participation
Time Frame: 3months
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Pediatric Aquatic Therapy: *Children diagnosed with CP, spastic type,*4 to 12 years of age,*Goss Motor Functional Classification System (GMFCS) level I-IV, participate pediatric aquatic therapy according preference
- Conventional Therapy: Children diagnosed with CP, spastic type,*4 to 12 years of age,*Goss Motor Functional Classification System (GMFCS) level I-IV, participate conventional therapy according preference
Arm/Group | Pediatric Aquatic Therapy | Conventional Therapy
Number analyzed (Participants) | 11 | 13
units on a scale | 69.6 (8.3) | 68.5 (14.6)
Statistical Analysis 1: Comparison: Pediatric Aquatic Therapy vs Conventional Therapy; null hypothesis : there is no difference in social participation between pediatric aquatic therapy group and conventional therapy group; Test type: Superiority or Other; p = 0.332, ANCOVA

ADVERSE EVENTS:
Time Frame: 3 months
Description: no pain or falling down or other adverse effect were report
Groups:
- Effects of Pediatric Aquatic Therapy on Motor Performance: *Children diagnosed with CP, spastic type,*4 to 12 years of age,*Goss Motor Functional Classification System (GMFCS) level I-IV,
Arm/Group | Effects of Pediatric Aquatic Therapy on Motor Performance
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
no pain or falling down or other adverse effect were report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less